CLINICAL TRIAL: NCT04126187
Title: AcrySof® Bilateral PanOptix(R) Spectacle Freedom and Patient Satisfaction Study
Status: Completed | Type: Observational
Sponsor: Gainesville Eye Associates (Other)
Collaborators: Science in Vision (Other)
Responsible Party: Sponsor
Other Study IDs: CB-19-002
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Results first posted 2021-08-11 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Cataract
Keywords: Panoptix; Trifocal IOL; Multifocal IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Panoptix: Bilateral implantation of the Panoptix trifocal IOL
  Interventions: Device: Panoptix

INTERVENTIONS:
Device: Panoptix — Panoptix trifocal intraocular lens (IOL)

SUMMARY:
The objective of this study is to assess the spectacle independence of patients receiving the AcrySof® Panoptix® Intraocular lens (IOL) after uneventful cataract surgery.

DETAILED DESCRIPTION:
This study is a single-arm unmasked clinical evaluation study of spectacle independence after successful bilateral cataract surgery. Subjects will be assessed pre-operatively, operatively and at 1 day, 1 month and 3 months post-operatively. Clinical evaluations will include administration of a spectacle independence questionnaire, as well as measurement of bilateral visual acuity and manifest refraction.

ELIGIBILITY:
Inclusion Criteria

Subjects are eligible for the study if they meet the following criteria:

Note: Ocular criteria must be met in both eyes.

* Presenting for uncomplicated bilateral cataract surgery and have an interest in spectacle independence using a multifocal IOL or multifocal toric IOL option
* Gender: Males and Females.
* Age: 40 or older.
* Willing and able to provide written informed consent for participation in the study.
* Willing and able to comply with scheduled visits and other study procedures.
* Have good ocular health, with no pathology that compromises visual acuity (outside of residual refractive error and cataract)
* Have regular corneal astigmatism with a magnitude that can be treated with a non-toric IOL or a toric IOL in the approved ranged for the Panoptix lens.
* Have 20/32 (0.2 logMAR) or better potential acuity in both eyes

Exclusion Criteria If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Irregular astigmatism (e.g. keratoconus)
* Corneal pathology (e.g. scar, dystrophy, pterygium, moderate-to-severe dry eye)
* Monocular status (e.g. amblyopia)
* Previous radial keratotomy, corneal refractive surgery or other corneal surgery (e.g. corneal transplant, lamellar keratoplasty)
* Previous anterior or posterior chamber surgery (e.g., vitrectomy, laser iridotomy)
* Diabetic retinopathy
* Macular pathology (e.g. age-related macular degeneration, epiretinal membrane)
* History of retinal detachment
* Subjects who have an acute or chronic disease or illness that would confound the results of this investigation (e.g., immunocompromised, connective tissue disease, clinically significant atopic disease, diabetes, and any other such disease or illness), that are known to affect postoperative visual acuity.
* Participation in (or current participation) any investigational drug or device trial within the previous 30 days prior to the start date of this trial.

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects ≥40 years of age presenting for cataract surgery who are interested in spectacle lens freedom and considered appropriate candidates for multifocal lens implantation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clayton G Blehm, MD, Principal Investigator — Gainesville Eye Associates
Locations (1):
- Gainesville Eye Associates, Gainesville, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morlock R, Wirth RJ, Tally SR, Garufis C, Heichel CWD. Patient-Reported Spectacle Independence Questionnaire (PRSIQ): Development and Validation. Am J Ophthalmol. 2017 Jun;178:101-114. doi: 10.1016/j.ajo.2017.03.018. Epub 2017 Mar 22. PMID 28341605

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Panoptix
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Panoptix
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Have Spectacle Independence
Description: Percent of patients who never or rarely wear spectacles for distance, intermediate or near vision 3 months postop (based on the Patient-Reported Spectacle Independence Questionnaire (PRSIQ) - "a little of the time" or "none of the time")
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Panoptix
Number analyzed (Participants) | 30
Participants | 27

2. Secondary Outcome: Binocular Uncorrected Distance Visual Acuity
Description: Binocular uncorrected distance visual acuity in logMAR
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Panoptix
Number analyzed (Participants) | 30
logMAR | .09 (.09)

3. Secondary Outcome: Binocular Uncorrected Intermediate Visual Acuity
Description: Binocular uncorrected intermediate visual acuity in logMAR
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Panoptix
Number analyzed (Participants) | 30
logMAR | 0 (.1)

4. Secondary Outcome: Binocular Uncorrected Near Visual Acuity
Description: Binocular logMAR uncorrected near visual acuity
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Panoptix
Number analyzed (Participants) | 30
logMAR | .03 (.11)

5. Secondary Outcome: Binocular Best-corrected Distance Visual Acuity
Description: Binocular logMAR best-corrected distance visual acuity
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Panoptix
Number analyzed (Participants) | 30
logMAR | .02 (.05)

6. Secondary Outcome: Binocular Distance-corrected Intermediate Visual Acuity
Description: Binocular distance-corrected logMAR intermediate visual acuity
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Panoptix
Number analyzed (Participants) | 30
logMAR | -.02 (.09)

7. Secondary Outcome: Binocular Distance-corrected Near Visual Acuity
Description: Binocular logMAR distance-corrected near visual acuity
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Panoptix
Number analyzed (Participants) | 30
logMAR | -.01 (.07)

8. Secondary Outcome: Spherical Equivalent Refraction
Description: Spherical equivalent refraction in diopters
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Panoptix
Number analyzed (Participants) | 30
diopters | -.02 (.35)

9. Secondary Outcome: Residual Refractive Cylinder
Description: Residual refractive cylinder in diopters
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Panoptix
Number analyzed (Participants) | 30
diopters | 0.21 (.28)

10. Secondary Outcome: Number of Participants Who Are Spectacle Independent in the Emmetropia Subgroup
Description: Spectacle independence of subjects that hit refractive target within 0.5 diopters (D) spherical equivalent refraction
Time Frame: 3 months
Population: This is the number of patients that had a refractive target within 0.50D of intended (emmetropia subgroup)
Measure: Count of Participants; unit: Participants
Arm/Group | Panoptix
Number analyzed (Participants) | 22
Participants | 21

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Panoptix
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/87/NCT04126187/Prot_SAP_000.pdf